CLINICAL TRIAL: NCT06425341
Title: A Multicenter, Randomized, Open, Parallel-designed Phase II Study to Evaluate the Efficacy and Safety of HRS-5635 Injection Alone or in Combination With Other Agents in Patients Treated for Chronic Hepatitis B
Brief Title: A Multicenter, Randomized, Open, Parallel-designed Study to Evaluate the Efficacy and Safety of HRS-5635 Injection Alone or in Combination With Other Agents in Patients Treated for Chronic Hepatitis B
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-5635-201
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-07

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Intervention Model Description: Multi-center, random, open, parallel design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- HRS-5635 Injection dose 1 (Experimental)
  Interventions: Drug: HRS-5635 Injection
- HRS-5635 Injection dose 2 (Experimental)
  Interventions: Drug: HRS-5635 Injection
- HRS-5635 Injection dose 3 (Experimental)
  Interventions: Drug: HRS-5635 Injection
- HRS-5635 Injection dose 4 (Experimental)
  Interventions: Drug: HRS-5635 Injection
- HRS-5635 Injection (low dose) and Peg-IFN-α, administered by subcutaneous injection (Experimental)
  Interventions: Drug: HRS-5635 Injection (low dose) and Peg-IFN-α
- HRS-5635 Injection (high dose) and Peg-IFN-α, administered by subcutaneous injection (Experimental)
  Interventions: Drug: HRS-5635 Injection (high dose) and Peg-IFN-α
- Peg-IFN-α, administered by subcutaneous injection (Placebo Comparator)
  Interventions: Drug: Peg-IFN-α
- HRS-5635 Injection with Peg-IFN-α（Part C） (Experimental)
  Interventions: Drug: HRS-5635 Injection with Peg-IFN-α
- HRS-5635 Injection（Part D） (Experimental)
  Interventions: Drug: HRS-5635 Injection

INTERVENTIONS:
Drug: HRS-5635 Injection — HRS-5635 Injection low dose administered by subcutaneous injection
  Arms: HRS-5635 Injection dose 1
Drug: HRS-5635 Injection — HRS-5635 Injection medium dose administered by subcutaneous injection
  Arms: HRS-5635 Injection dose 2
Drug: HRS-5635 Injection — HRS-5635 Injection high dose administered by subcutaneous injection
  Arms: HRS-5635 Injection dose 3
Drug: HRS-5635 Injection — HRS-5635 Injection lowest dose administered by subcutaneous injection
  Arms: HRS-5635 Injection dose 4
Drug: HRS-5635 Injection (low dose) and Peg-IFN-α — HRS-5635 Injection (low dose) and Peg-IFN-α, administered by subcutaneous injection
  Arms: HRS-5635 Injection (low dose) and Peg-IFN-α, administered by subcutaneous injection
Drug: HRS-5635 Injection (high dose) and Peg-IFN-α — HRS-5635 Injection (high dose) and Peg-IFN-α, administered by subcutaneous injection
  Arms: HRS-5635 Injection (high dose) and Peg-IFN-α, administered by subcutaneous injection
Drug: Peg-IFN-α — Peg-IFN-α, administered by subcutaneous injection
  Arms: Peg-IFN-α, administered by subcutaneous injection
Drug: HRS-5635 Injection with Peg-IFN-α — HRS-5635 Injection and Peg-IFN-α, administered by subcutaneous injection
  Arms: HRS-5635 Injection with Peg-IFN-α（Part C）
Drug: HRS-5635 Injection — HRS-5635 Injection, administered by subcutaneous injection
  Arms: HRS-5635 Injection（Part D）

SUMMARY:
A multicenter, randomized, open, parallel-designed Phase II study to evaluate the efficacy and safety of HRS-5635 injection alone or in combination with other agents in patients treated for chronic hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the body mass index standard greater than or equal to 18.5 kg/m2 and less than 35 kg/m2;
2. Chronic hepatitis B defined as HBV infection documented for at least 6 months prior to screening;
3. Virologically suppressed on nucleoside or nucleotide analogues treatment with HBV DNA below the lower limit of quantitation;
4. On commercially available NAs monotherapy for at least 24 weeks before randomization, and the dosing regimen remained unchanged for at least 4 weeks before randomization;
5. Need to take effective contraceptive measures；
6. Volunteer to sign an informed consent.

Exclusion Criteria:

1. History of cirrhosis or clinical evidence of hepatic decompensation, confirmed or suspected liver cancer, with other liver diseases other than chronic hepatitis B that may affect the evaluation of the study;
2. With autoimmune disease;
3. History of solid organ transplantation or hematopoietic stem cell transplantation;
4. Clinically significant and unstable or uncontrolled severe cardiovascular and cerebrovascular diseases;
5. Malignant tumors were diagnosed within 5 years prior to randomization；
6. Infection requiring intervention within 2 weeks prior to randomization;
7. Major trauma or major surgery within the 12 weeks prior to randomization, or surgical plans or other treatment during the study period which the investigators determined may influence the evaluation of the study results;
8. Laboratory tests during the screening period were obviously abnormal;
9. Prolonged ECG QTcF or other clinically significant abnormal results that may pose a significant safety risk to the subject during the screening period;
10. History of drug use, alcohol or drug abuse in the 12 months prior to randomization;
11. Participated in clinical study of other drugs (received experimental drugs);
12. Pregnant or nursing women;
13. Allergic to a drug ingredient or component;
14. Other reasons for ineligibility as judged by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 369 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-01-19 (Estimated)

PRIMARY OUTCOMES:
PartA：Change in mean log10 serum hepatitis B surface antigen levels from baseline at week 12 | Week 12
PartB：Proportion of subjects whose serum hepatitis B surface antigen (HBsAg) had turned negative at week 48 | Week 48
PartC：Proportion of subjects whose serum hepatitis B surface antigen (HBsAg) had turned negative at week 48 | Week 48
PartD：Proportion of subjects whose serum hepatitis B surface antigen (HBsAg) had turned negative at week 48 | Week 48

SECONDARY OUTCOMES:
Changes from baseline in mean log10 serum hepatitis B surface antigen levels | Pre-specified time points up to 72 weeks
Proportion of subjects with at least one log10 decline from baseline in serum hepatitis B surface antigen | Pre-specified time points up to 72 weeks
Proportion of subjects with serum hepatitis B surface antigen loss | Pre-specified time points up to 72 weeks
Proportion of subjects with serum hepatitis B surface antigen seroconversion | Pre-specified time points up to 72 weeks
Proportion of subjects with hepatitis B e-antigen loss | Pre-specified time points up to 72 weeks
Proportion of subjects with serum hepatitis B e-antigen seroconversion | Pre-specified time points up to 72 weeks
Proportion of subjects with virologic breakthrough | Pre-specified time points up to 72 weeks
Proportion of subjects with drug resistance | Pre-specified time points up to 72 weeks
Proportion of subjects who meet the criteria for stopping NA therapy | From 48 weeks to 72 weeks
Proportion of subjects with serum hepatitis B surface antigen loss and HBV DNA loss | Week 48

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided